CLINICAL TRIAL: NCT01471405
Title: Retrospective Non-interventional Study Evaluating Treatment Adaption During a One Year Follow-up After Completion of the 2-79-52030-207 Study in a Group of Acromegalic Patients With Macroadenoma Who Received 12 Injections of Lanreotide Autogel® 120 mg
Brief Title: One Year Follow-up of Study 2-79-52030-207 (PRIMARYS) in Acromegalic Patients With Macroadenoma
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: 8-79-52030-742
Record Dates: First submitted 2011-11-10; First posted 2011-11-15 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This non-interventional retrospective study aims to describe the therapeutic procedures and modalities received by patients and the correlation to hormone status, during a one year follow up from completion of the 2-79-52030-207 study.

ELIGIBILITY:
Inclusion Criteria:

* Completed the 2-79-52030-207 study and received 12 injections of lanreotide Autogel 120 mg, regardless of efficacy at the end of this period.
* Subject or in case of subject's death next of kin having given their written informed consent prior to collection of the data by the sponsor (if locally required)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients maintained on medical treatment with lanreotide Autogel | 1 year
Proportion of patients receiving other medical treatments | 1 year

SECONDARY OUTCOMES:
Proportion of patients with at least one pituitary surgery | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (18):
- III. Interní klinika Karlova Univerzita, Prague, Czechia
- France (9):
  - CHU de Rouen, Bois-Guillaume
  - Groupement hôspitalier est Federation d'endocrinologie., Bron
  - CHU Michallon, Grenoble
  - Hôpital Claude Huriez, Lille
  - CHU Timone, Marseille
  - Hôpital Bicêtre, Paris
  - Hôpital Haut Leveque, Pessac
  - CHU de Reims, Reims
  - Hôpital Larrey, Toulouse
- Germany (2):
  - Universität Duisburg-Essen, Essen
  - Klinikum der Johann Wolfgang, Goethe-Universität, Frankfurt
- Italy (2):
  - Università Federico II di Napoli, Napoli
  - Università Cattolica del Sacro Cuore, Roma
- İstanbul Universitesi, Cerrahpaşa Tıp Fakültesi, Istanbul, Turkey (Türkiye)
- United Kingdom (3):
  - Aberdeen Royal Infirmary, Aberdeen
  - Christie Hospital, Manchester
  - Derriford Hospital, Plymouth

REFERENCES:
- See also: 2-79-52030-207 (NCT00690898) — http://clinicaltrials.gov/ct2/show/NCT00690898?term=2-79-52030-207&rank=1